CLINICAL TRIAL: NCT00350831
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of the KIT Inhibitor XL820 Administered Orally Daily to Subjects With Solid Tumors
Brief Title: Study of XL820 Given Orally Daily to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL820-002
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Cancer
Keywords: Solid tumor
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: XL820

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the KIT inhibitor XL820 when given orally daily to adults with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a histologically confirmed solid tumor that is metastatic or unresectable for which known effective measures do not exist or are no longer effective, and there are no known therapies to prolong survival
* Subject is at least 18 years old
* Subject has ECOG performance status ≤ 2
* Subject has a life expectancy of > 3 months
* Subject has adequate organ and marrow function
* In the adrenocorticotropic hormone (ACTH) stimulation test, the subject has a serum cortisol level ≥ 20 ug/dL (552 nmol/L) 30-90 minutes after injection of ACTH
* Subject has given written informed consent
* Sexually active subjects (male and female) must use accepted methods of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* Subject has received anticancer treatment within 30 days before the first dose of XL820, or has not recovered to grade ≤ 1 from adverse events due to agents administered more than 30 days earlier
* Subject has received radiation to ≥ 25% of his/her bone marrow within 30 days of XL820 treatment
* Subject has received an investigational agent within 30 days of the first dose of XL820
* Subject has known brain metastases
* Subject has known uncontrolled intercurrent illness
* Subject is pregnant or lactating
* Subject is known to be positive for HIV
* Subject has a known allergy or hypersensitivity to any of the components of the XL820 formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-07

PRIMARY OUTCOMES:
maximum tolerated dose
safety and tolerability

SECONDARY OUTCOMES:
plasma pharmacokinetics
pharmacodynamic effects
long-term safety and tolerability

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cancer Therapy and Research Center, San Antonio, Texas